CLINICAL TRIAL: NCT01369186
Title: Drug Drug Interactions of Antiplatelet Drugs and Morphine
Brief Title: Drug Drug Interactions of Aspirin and P2Y12-inhibitors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Eva-Luise Hobl, Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-023761-22
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Drug Interaction Potentiation; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Morphine; vendal neu

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Active Comparator): Vendal 5 mg i.v. bolus injection
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator): Sodium chloride 0.9% i.v. bolus injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine — i.v. bolus injection
  Other Names: Vendal
  Arms: Morphine
Drug: Placebo — i.v. bolus injection
  Other Names: Sodium chloride 0,9%
  Arms: Placebo

SUMMARY:
Study Objective: To investigate potential drug-drug interactions (pharmacokinetics and pharmacodynamics) of morphine and antiplatelet drugs (aspirin, clopidogrel, prasugrel, ticagrelor)

DETAILED DESCRIPTION:
Rationale: Opiates reduce the intestinal resorption of orally administered drugs such as paracetamol. Because morphine is often injected to relieve pain in patients with myocardial infarction, it is of particular interest if morphine may decrease the rate of absorption of antiplatelet drugs. Results of this study will provide essential information for the use of morphine and antiplatelet drugs in clinical practice, in particular in myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ≥ 18 years of age
* No intake of NSARs and P2Y12-inhibitors within 14 days before study entry
* Written informed consent

Exclusion Criteria:

* Known coagulation disorders
* Relevant impairment of hepatic function (elevated transaminases, ≥ 2 fold)
* Relevant impairment of renal function
* Infectious diseases (HIV, hepatitis B and C)
* Gestation and lactation
* Clinically relevant abnormal laboratory values
* Use of medication during 2 weeks before the start of the study, which may affect the validity of the study
* General contraindications for aspirin (resp. clopidogrel, prasugrel, ticagrelor) and morphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Platelet function | 14 days

SECONDARY OUTCOMES:
Tmax | 14 days
Cmax | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

REFERENCES:
- [Background] Hobl EL, Schmid RW, Stimpfl T, Ebner J, Jilma B. Absorption kinetics of low-dose chewable aspirin--implications for acute coronary syndromes. Eur J Clin Invest. 2015 Jan;45(1):13-7. doi: 10.1111/eci.12373. PMID 25402445
- [Background] Hobl EL, Stimpfl T, Ebner J, Schoergenhofer C, Derhaschnig U, Sunder-Plassmann R, Jilma-Stohlawetz P, Mannhalter C, Posch M, Jilma B. Morphine decreases clopidogrel concentrations and effects: a randomized, double-blind, placebo-controlled trial. J Am Coll Cardiol. 2014 Feb 25;63(7):630-635. doi: 10.1016/j.jacc.2013.10.068. Epub 2013 Dec 4. PMID 24315907
- [Derived] Hobl EL, Reiter B, Schoergenhofer C, Schwameis M, Derhaschnig U, Lang IM, Stimpfl T, Jilma B. Morphine interaction with prasugrel: a double-blind, cross-over trial in healthy volunteers. Clin Res Cardiol. 2016 Apr;105(4):349-55. doi: 10.1007/s00392-015-0927-z. Epub 2015 Oct 22. PMID 26493304